CLINICAL TRIAL: NCT02208739
Title: Effect of Nonsurgical Periodontal Therapy Verses Oral Hygiene Instructions on Clinical Parameters as Well as Immunological and Microbial Profile of Patients With Chronic Periodontitis
Brief Title: Effect of Nonsurgical Periodontal Therapy Verses Oral Hygiene Instructions on Patients With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPPC-C2
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; periodontal pathogens; inflammatory mediators; Non surgical periodontal therapy; Oral hygiene instructions; Polymerase chain reaction; Elisa
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nonsurgical periodontal therapy (Experimental): Nonsurgical periodontal therapy was given to all patients at baseline
  Interventions: Procedure: Nonsurgical periodontal therapy
- Oral hygiene instructions (Active Comparator): Oral hygiene instructions were given to all patients at baseline
  Interventions: Procedure: Nonsurgical periodontal therapy; Procedure: Oral hygiene instructions

INTERVENTIONS:
Procedure: Nonsurgical periodontal therapy — All patients were instructed in oral hygiene methods using a soft bristled toothbrush, a compact-tuft toothbrush, interdental brushes and dental floss utilizing the modified Bass technique. Full mouth debridement, which consisted of scaling and root planing, was done in a single visit for all subjects using an ultrasonic scaler and gracey curettes. Additionally, all patients were given a 0.12% Chlorhexidine mouthrinse (Hexipro®). They were instructed to rinse three times a day using 15ml each time for a period of 14 days commencing immediately after completion of full mouth debridement. Thereafter at each recall visit, all participants were re-motivated and professional prophylaxis was performed.
Procedure: Oral hygiene instructions — All patients were instructed in oral hygiene methods using a soft bristled toothbrush, a compact-tuft toothbrush, interdental brushes and dental floss utilizing the modified Bass technique.
  Arms: Oral hygiene instructions

SUMMARY:
Periodontitis, a bacterial dental biofilm based infectious disease, is a chronic inflammatory disease of the periodontium which results in irreversible destruction of supporting structures of the teeth such as periodontal ligaments, connective tissues, cementum and alveolar bone. More than 700 species of bacteria are estimated to be found in the sub-gingival dental biofilm in which periodontopathogens are found to be responsible in initiating periodontal disease. Chronic periodontitis, although termed as 'chronic', starts as an acute inflammation. Low levels of bacteremia and endotoxins provides a stimulus for the systemic inflammatory response. In periodontitis, the interaction of lipopolysaccharide (LPS) from gram-negative bacteria with host cells initiates the secretion of cytokines and the expression of cell adhesion molecules in gingival tissue which leads to loss of alveolar bone and connective tissues supporting the teeth.

In the management of chronic periodontitis, non surgical periodontal therapy (NSPT) which includes oral hygiene instruction (OHI), scaling and root planing, is administered to improve clinical parameters as well as controlling the bacterial count responsible in initiating the disease and the resultant inflammatory response. Success of the treatment can be analyzed when the clinical parameters, counts of the microbes is reduced and inflammatory response is controlled. Studies which have evaluated the microbiological and immunological response following NSPT clearly demonstrates an improvement in clinical parameters, reduction in inflammatory mediators present as well as a decrease in microbial count.

OHI which includes tooth brushing and inter-dental cleaning is found beneficial in removing microbial plaque, thus, preventing periodontal diseases such as gingivitis and periodontitis. Studies have evaluated the role of OHI on clinical and immunological parameters and microbiological profiles of periodontal maintenance subjects, while none of them evaluated its role alone in the management of chronic periodontitis subjects. Therefore, the purpose of the following investigation was to compare the changes in the clinical parameters, inflammatory mediators as well as level and frequency of detection of periodontopathogens that take place after 3-months of NSPT versus OHI and to evaluate if clinical parameters have an effect on these inflammatory mediators and microbiological changes.

DETAILED DESCRIPTION:
Subjects with moderate to advanced chronic periodontitis were selected for this longitudinal randomized clinical trial. Ethical clearance for the study was granted by the Medical Ethics Committee, Faculty of Dentistry, University of Malaya [Medical Ethics Committee Number: DF PE1002/0045(P)]. The study was conducted in accordance with the Helsinki Declaration of 1975, as revised in 2000. The CONSORT guidelines for clinical trials were followed.

Out of 112 screened patients 56 patients fulfilled the inclusion and exclusion criteria. Inclusion criteria were minimum of 12 teeth present with pocket of 5mm or more and probing attachment loss of 4mm or more in at least 2 different quadrants which bled on probing. Exclusion criteria included history of cardiovascular problems, pregnancy, smokers, and subjects receiving antibiotics in past 4 months or NSPT in past 6 months. Recruited patients were treated at the Periodontology clinic, Faculty of Dentistry, University of Malaya. Using Cohen's d formula it was calculated that at least 26 patients would be needed per treatment group to detect this difference with 80% power.

Prior to baseline examination, patients were assigned in the NSPT and OHI group using block randomization. Patients in NSPT group received OHI, scaling and root planing followed by 0.12% Chlorhexidine mouth rinses while patients in OHI group received OHI only. At each month recall visit, participants in both groups were reviewed and motivated. Professional prophylaxis was only received by NSPT group. Two calibrated examiners (RPCR and WNAWA) performed all treatment on the patients. Probing pocket depth ( PPD), probing attachment loss (PAL), gingival bleeding index (BI) and visible plaque index (PI) were determined on all present teeth except third molars at baseline and 3 months after therapy. For PI and BI, 4 sites were measured (mesial, distal, buccal, lingual) and for PPD and PAL 6 sites were recorded (disto-buccal, mid-buccal, mesio-buccal, mesio-lingual, mid-lingual and disto-lingual). Utilizing Kappa statistics, good agreements (>0.8) were obtained for intra and inter operator reproducibility of all recorded clinical parameters.

Identification of subgingival microbiota using quantitative polymerase chain reaction technique.

Sub-gingival plaque scraping samples were obtained at baseline and 3-months post therapy with sterile curettes from the deepest sites at each quadrant and were pooled together for each subject. Prior to sampling, isolation was maintained with cotton rolls and supra-gingival plaque was removed using cotton pellets. Plaque scrapings were re-suspended in 1.5 ml of Phosphate Buffered Saline and stored at -80⁰C freezer prior to DNA extraction. 100µl of plaque sample was used for automated DNA extraction in the lab using the Qiacube machine (Qiagen®, Biotechnology, Netherlands). The tubes containing the plaque samples were centrifuged at a speed of 5,000 × g for 10 minutes on a tabletop centrifuge machine to obtain the pellet. The pellet was then used for automated DNA extraction with the Qiacube machine. 100µl of eluted DNA was stored in -20⁰C for bacterial detection using quantitative polymerase chain reaction (Applied Biosystem, USA).

Reference bacterial strains used in this study were P.gingivalis (W83), A.actinomycetemcomitans (NCTC9710), P.intermedia (ATCC25611) and T.forsythia (CCUG 21028AT). All the bacterial strains were grown as recommended by American Type Culture Collection (ATCC). After the growth of bacteria till late exponential phase they were washed with sterile distilled water and DNA extraction was carried out using the same protocol as for plaque samples.

The concentration and purity of extracted DNA was determined using spectrophotometer machine (Nanodrop 2000, Thermo scientific, USA). DNA concentration from both plaque samples and reference strain were calculated and recorded accordingly. The extracted DNAs were stored in -20⁰C until the initiation of quantitative polymerase chain reaction procedure.

The protocol given by Boutaga et al., (2005) was followed for quantitative polymerase chain reaction . Primers and probes selected for this study are shown in Table 1. A total reaction mixture of 20ul was used for amplification, which contains 2ul of template DNA from plaque sample/reference strain,10 ul of 2 x TaqMan fast advanced master mix (Applied biosystems, USA), 1ul of 20x gene expression assay and 7ul nuclease free water. All the components of reaction mixture except for DNA sample were added in 1.5ml micro centrifuge tube. The tube was vortexed and than centrifuged to eliminate air bubbles. Mixture was transferred to 96-well plate with addition of 2ul DNA sample. The Plate was then covered with optical adhesive and centrifuged again to make sure air bubbles are eliminated. The cycling conditions used were as follows: 50oc for 2min and 95oc for 10min followed by 45 cycles at 95oc for 15s and 60oc for 1min.

Dilutions of known amounts of reference strains of DNA were used to generate standard curves with correlation coefficient (R2: 0.99). For quantification/copy number determination, the results from unknown samples were projected on the standard curves obtained from the pure cultures using the formula: Quantity DNA=10(ct-b)/m.

Determination of Interleukin-1, Interleukin-6, Adiponectin and Tumour Necrosis Factor-alpha level in Serum.

All reagents were allowed to reach room temperature before use and were gently mixed prior to the experiments. Number of 8-well strips needed for the assay was determined. 100 ul of the Standard Diluent Buffer were added to zero wells and 1 well was reserved for chromogen blank. 100 ul of standards, samples and controls were added to the appropriate microtiter wells. 50 ul of biotinylated anti-Interleukin-6 (Biotin Conjugate) solution were pipetted into each well except the chromagen blank and then gently tapped on the side of the plate to mix. Next, plates were covered with plate covers and incubated for 2 hours at room temperature. Solutions were thoroughly aspirated from wells and the liquid discarded. The wells were washed 4 times. 100 ul streptavidin-histidine-rich protein working solution were added to each well except the chromogen blank. Again, the plates were covered with the plate covers and incubated for 30 minutes at room temperature. Solution from wells was thoroughly aspirated and the liquid discarded. The wells were washed 4 times. 100ul of Stabilized Chromogen was added to each well. The plates were incubated for 30 minutes at room temperature in the dark. 100 ul of stop solution was added to each well and then gently tapped on the side of the plate to mix. The absorbance of each well was read at 450 nm having blanked the plate reader against a chromogen blank composed of 100 ul each of Stabilized Chromogen and Stop Solution. The absorbance of the standards against the standard concentration was then plotted on graph paper.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have at least 12 teeth present
* Patients with Moderate to Advanced Chronic periodontitis
* Patients with 2 or more interproximal sites (not on same tooth) with probing pocket depths of 5mm or more and 2 or more interproximal sites (not on same tooth)of probing attachment loss of 4mm or more which bled on probing.

Exclusion Criteria:

* Patients who had history of systemic antibiotic usage over the previous 4 months
* Patients who were pregnant
* Patients who had received non-surgical periodontal treatment within the past 6 months
* Patients who had received surgical periodontal treatment within the past 12 months
* Patients who were smokers
* Patients with a history of stroke or an acute cardiovascular event over the previous 12 months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Effect of NSPT vs OHI on probing pocket depth of subjects with chronic periodontitis | Baseline to 3 months
  Outcome measurements assessed are probing pocket depth

SECONDARY OUTCOMES:
Effect of NSPT vs OHI on microbiological parameters of subjects with chronic periodontitis | Baseline to 3 months
  Changes in subgingival microbiota were assessed as changes in frequency of detection and microbial count of A.actinomycetemcomitans, T.forsythia, P.gingivalis and P.intermedia from baseline to 3 months post therapy.
Effect of NSPT vs OHI on immunological parameters of subjects with chronic periodontitis | Baseline to 3 months
  Changes in immunological parameters were assessed as changes in levels of high-sensitivity C-reactive protein , Interleukin-1, Interleukin-6. Tumour Necrosis Factor alpha, adiponectin and resistin from baseline to 3 months post therapy.
Effect of NSPT vs OHI on oral health related quality of life of subjects with chronic periodontitis | Baseline to 3 months
  Changes in oral health related quality of life from baseline to 3 months post therapy in both treatment groups.
Effect of NSPT vs OHI on plaque index of subjects with chronic periodontitis | Baseline to 3 months
  Outcome measurements assessed are Plaque index
Effect of NSPT vs OHI on gingival bleeding index of subjects with chronic periodontitis | Baseline to 3 months
  Outcome measurements assessed are Gingival bleeding index
Effect of NSPT vs OHI on clinical attachment level of subjects with chronic periodontitis | Baseline to 3 months
  Outcome measurements assessed are clinical attachment levels
Effect of NSPT vs OHI on oral health related quality of life of subjects with chronic periodontitis | Baseline to 3 months
  Outcome measurements assessed are oral health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Rathna D Vaithilingam, MClinDent, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Doungudomdacha S, Rawlinson A, Walsh TF, Douglas CW. Effect of non-surgical periodontal treatment on clinical parameters and the numbers of Porphyromonas gingivalis, Prevotella intermedia and Actinobacillus actinomycetemcomitans at adult periodontitis sites. J Clin Periodontol. 2001 May;28(5):437-45. doi: 10.1034/j.1600-051x.2001.028005437.x. PMID 11350507
- [Background] Knofler GU, Purschwitz RE, Eick S, Pfister W, Roedel M, Jentsch HF. Microbiologic findings 1 year after partial- and full-mouth scaling in the treatment of moderate chronic periodontitis. Quintessence Int. 2011 Oct;42(9):e107-17. PMID 21909493